CLINICAL TRIAL: NCT04012528
Title: Assesment of Enhanced Recovery After Pediatric Idiopathic Scoliosis Surgery
Brief Title: ERAS and Pediatric Scoliosis Surgery
Acronym: RAAC
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: RECHMPL18_0382
Record Dates: First submitted 2019-04-26; First posted 2019-07-09 (Actual); Last update posted 2020-12-29 (Actual); Status verified 2020-12

CONDITIONS: Scoliosis
Keywords: Pediatric; Surgery; Rehabilitation
MeSH Terms: conditions — Scoliosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- "the before" group: 75 teenagers after scoliosis surgery before ERAS program implementation
  Interventions: Other: ERAS program
- "the after" group: 75 teenagers after scoliosis surgery after ERAS program implementation

INTERVENTIONS:
Other: ERAS program — ERAS program
  Groups: "the before" group

SUMMARY:
The aim of this study is to compare the outcomes after scoliosis surgery before and after ERAS (enhanced recovery after surgery) program inplementation in children and teenager.

DETAILED DESCRIPTION:
Enhanced recovery after surgery (ERAS) is a multimodal approach focused on reducing the stress response and associated physiologic changes related to surgery. Over the past 20 years, ERAS programs have been found to result in reduced lenght of stay and complications in adult patients. Data in pediatric population remains very scarce.Therefore this study was designed to compare the outcomes after scoliosis surgery before and after ERAS (enhanced recovery after surgery) program inplementation in children and teenager.

ELIGIBILITY:
Inclusion criteria:

* patient with age < 18 years
* patient scheduled for scoliosis surgery

Exclusion criteria:

* patient with age > 18years
* patient with medical follow up by pediatric chronic pain departement

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Chidren and teenager admitted for scoliosis surgery
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-11-01 (Actual); Study Completion 2021-11-30 (Estimated)

PRIMARY OUTCOMES:
Postoperative length of hospital stay | up to 4 weeks after surgery
  Postoperative length of hospital stay

SECONDARY OUTCOMES:
Number of Antalgics consumption | up to 15 days after surgery
  Antalgics consumption including opioids and non-opioids drug
Time to oral diet tolerance | up to 15 days after surgery
  Able to eat without abdominal discomfort, nausea, or vomiting
Time to first bowel motion | up to 15 days after surgery
  Able to eat without abdominal discomfort, nausea, or vomiting
Time to first verticalization | up to 15 days after surgery
  Able to eat without abdominal discomfort, nausea, or vomiting

CONTACTS AND LOCATIONS:
Overall Officials: Chrystelle CS SOLA, MD, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Uh Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: Undecided
NC